CLINICAL TRIAL: NCT06828302
Title: Internet-delivered Parent-Child Interaction for Parents of Children 2-7 Years With Disruptive Behaviors
Acronym: iPCIT pilot
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Marianne Bonnert, PhD, lic psych, principal investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPM Dnr: 2024-06544-01
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-10

CONDITIONS: Disruptive Behavior
Keywords: Internet-CBT; Parent; Children; Parent-Child Interaction Therapy
MeSH Terms: conditions — Problem Behavior

STUDY DESIGN:
Intervention Model Description: Uncontrolled feasibility study using pretest-posttest design with 2 mo FU as primary endpoint.
Masking Description: Self-reported outcomes assessed online without any influence from study staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iPCIT (Other): Online parent management training (PMT) to teach parental skills (10 weekly online modules) combined with videosession for coaching of parental skills (5 biweekly sessions)
  Interventions: Behavioral: Internet-delivered Parent-Child Interaction Therapy

INTERVENTIONS:
Behavioral: Internet-delivered Parent-Child Interaction Therapy — Parent management training delivered online where Internet-modules are combined with video sessions for live coaching.
  Other Names: Internet-CBT; Internet-delivered cognitive behavior therapy

SUMMARY:
The goal of this feasibility study is to evaluate feasibility of Internet-delivered Parent-Child Interaction Therapy for parents of children 2-7 years with disruptive behaviors. The main questions it aims to answer are:

1. Could a brief online version of PCIT (iPCIT) be feasible for reducing disruptive behaviors and internalizing problems in young children, and for improving the quality of parent-child interaction?
2. How is iPCIT experienced by participating parents?

Participants will receive a 10-week online intervention of Parent-Child Interaction Therapy and answer questionnaires online weekly.

DETAILED DESCRIPTION:
Severe early behavioral problems increase the risk of impaired functioning in childhood and later life. Parent-Child Interaction Therapy (PCIT) is particularly effective for young children (age 2-7) with disruptive behaviors but is unimplemented in Sweden. Barriers to PCIT implementation include time constraints for parents and therapist challenges. An abbreviated internet-delivered version, iPCIT, may address these barriers. The objective of the study is to evaluate feasibility and acceptability of iPCIT.

Research questions

This study will use an uncontrolled pretest-posttest design, all participants will receive the intervention. The intervention consists of 10 weekly modules delivered over the Internet with guided support from an experienced CBT-trained psychologist and 5 biweekly videosessions where parents practice parental skills in a play situation with their child while receiving feedback and support from their therapist.

Assessments will be made pretreatment, weekly during treatment for the primary outcome and potential mediators, posttreatment, at the primary endpoint 2 months after treatment completion and at follow up 6 months after treatment completion. Twenty participants (parents of children aged 2-7 years) will be included. All outcome data will be collected digitally and include for feasibility: treatment credibility, working alliance, compliance with the treatment (number of modules completed), any adverse events, subjective overall relief and satisfaction with treatment. For potential efficacy, the clinical effect in the group will be analyzed on pre- to post-measurements, including weekly measurements and 2 months follow up after treatment termination (primary endpoint). The participants will be followed 6 months after treatment completion to analyze long term clinical effects.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-7 years
* Disruptive behaviors as assessed with Eyberg Child Behavior Inventory (ECBI) ≥126 for boys and ≥121 for girls (which corresponds to the 90th percentile according to Swedish norms)
* Language ability equivalent to at least an average 2-year-old, defined as a vocabulary of ≥ 25 word and ability to understand simple instructions, assessed with a language screening form

Exclusion Criteria:

* Severe autism spectrum condition (autism level 2 or 3 or equivalent functioning)
* parents who are not proficient enough in the Swedish language to complete questionnaries and receive therapy without an interpreter
* Presence of severe parental psychiatric disorders such as psychosis or suicidal ideations
* Ongoing severe psychosocial distress such as custody dispute.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Eyberg Child Behavior Inventory | From pretreatment to 18 weeks
  Caregiver report form measuring disruptive behaviors in children. 36 items with answers ranging from 1 (never) to 7 (always). Minimum value: 36. Maximum value: 252. A higher score means worse outcome.

SECONDARY OUTCOMES:
Weekly assessment of Child Behavior Forms | From pretreatment to 18 weeks
  Short caregiver report form measuring disruptive behaviors in children. Two scales with 9 items each with answers ranging from 1 (never) to 7 (always). Minimum value: 9. Maximum value: 63. A higher score means worse outcome.
Child Behavior Checklist | From pretreatment to 10 weeks
  Caregiver report form identifying problem behavior in children. 99 items with answers ranging from 0 (do not agree) to 2 (strongly agree). Minimum value: 0. Maximum value: 198. A higher score means worse outcome.
Dyadic Parent-Child Interaction Coding System | From pretreatment to 10 weeks
  Observation System measuring parental behavior and child behavior. The frequency of specified behaviors are measured during a five minute long standardized play situation.
Brunnsviken Brief Quality of Life Scale | From pretreatment to 18 weeks
  Questionnaire about quality of life. 12 items with answers ranging from 1 (strongly disagree) to 4 (strongly agree). Minimum value: 0. Maximum value: 96. A higher score means better outcome.
Perceived Stress Scale | From pretreatment to 18 weeks
  Questionnaire measuring overall stress. A 7-item version of the scale will be used with answers ranging from 0 (never) to 4 (very often). Minimum value: 0. Maximum value: 28. A higher score means worse outcome.
Parental Stress Scale | From pretreatment to 18 weeks
  Questionnaire measuring stress induced by parenthood. 18 items with answers from 1 ("strongly disagree") to 5 ("strongly agree"). Minimum value: 18. Maximum value: 90. A higher score means worse outcome.
Difficulties in Emotion Regulation Scale | From pretreatment to 18 weeks
  Questionnaire measuring emotion regulation ability. 16 items with answers ranging from 1 (almost never) to 5 (almost always). Minimum value: 16. Maximum value: 80. A higher score means worse outcome.
Parenting Young Children Scale | From pretreatment to 18 weeks
  Questionnaire measuring parental strategies. 6 items with answers ranging from 1 (never) to 7 (many times a day). Minimum value: 6. Maximum value: 42. A higher score means better outcome.

OTHER OUTCOMES:
Working Alliance Inventory | Treatment week 3
  Questionnaire measuring alliance with therapist. 6 items scored on a scale from 1 (never) to 7 (always). Minimum value: 6. Maximum value: 42. A higher score means better outcome.
Credibility Rating Scale | Treatment week 3
  Questionnaire measuring treatment credibility. 5 items scored on a scale from 0 (not at all) to 10 (very). Minimum value: 0. Maximum value: 50. A higher score means better outcome.
The Client Satisfaction Questionnaire | Posstreatment (treatment week 10)
  Questionnaire measuring satisfaction with treatment. 8 items with answers ranging from 1 (bad) to 4 (very good). Minimum value: 8. Maximum value: 32. A higher score means better outcome.
Subjective Adequate Relief Questionnaire | Posstreatment (treatment week 10)
  Questionnaire that measures self-perceived change in symptoms as a result of the treatment. The scale consists of 1 item rated from 0 (much worse) to 6 (much better).
Adverse events questionnaire | Posstreatment (treatment week 10)
  Short 6-item questionnaire to identify if any adverse events have occurred due to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Bonnert, PhD, Principal Investigator — Centre for Psychiatry Research, Karolinska Institutet & Stockholm Health Care Stockholm Sweden
Locations (1):
- Centre for Psychiatry Research, Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided